CLINICAL TRIAL: NCT06350396
Title: rTMS Intervention for DMPFC Treatment of Treatment-Resistant Depression Under the Guidance of Personalized Brain Functional Area Dissection (pBFS) Technology
Brief Title: pBFS-guided rTMS Over DMPFC for Treatment-Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLTRDDM2024
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
Keywords: Treatment Resistant Depression; Major Depression, Moderate Depression, MDD; personalized neuromodulation; Personalized Brain Functional Sectors
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS treatment (Experimental): 3 sessions of active rTMS would be delivered to the left DMPFC daily, with 1800 pulse/session.
  Interventions: Device: active rTMS treatment
- sham control (Sham Comparator): The identical treatment parameters will be administered akin to the active rTMS treatment, albeit devoid of actual stimulation.
  Interventions: Device: sham rTMS treatment

INTERVENTIONS:
Device: active rTMS treatment — Participants will receive 3 sessions per day of 1800 pulses per session, lasting for 21 days. Individualized targets will be generated using the pBFS method.
  Arms: active rTMS treatment
Device: sham rTMS treatment — The parameters in the sham arms are the same as the active stimulation groups. Stimulation was delivered by the same device as the active group fitted with a sham coil.
  Arms: sham control

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled trial aimed at exploring the effectiveness and safety of rTMS intervention with DMPFC targets guided by pBFS in patients with treatment-resistant depression.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established therapy for treatment-resistant depression. The dorsomedial prefrontal cortex (DMPFC), which serves as a connection intermediary of the aberrant functional network in cognitive control and rumination in depression, is highly correlated with disease manifestations and post-treatment improvements through several studies involving neuroimaging and brain injury. Research has shown that the response of DMPFC to rTMS is more subject to improving the dimensions of anxiety and insomnia in depression. Therefore, exploring the novel target DMPFC is also beneficial for distinguishing disease dimensions in the future, thereby enabling personalized treatment and improving clinical treatment efficacy.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized double-blind in a 1:1 ratio to the active rTMS group, or sham-control group. Then all participants will undergo a 21-day rTMS modulation and a 3-week, 9-week, and 6-month post-treatment follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients who meet the diagnostic criteria for depression in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and are not accompanied by psychiatric symptoms, with single or repeated episodes;
* (2) The Hamilton Depression Scale (HAMD) score for 17 items before randomization was ≥ 20 points, and the Montgomery Asberg Depression Rating Scale (MADRS) score was ≥ 20 points;
* (3) Individuals aged ≥ 18 and ≤ 65 years old, regardless of gender;
* (4) Currently, at least one antidepressant has been used for 6 weeks and the dosage used cannot be lower than the prescribed range of drug use;
* (5) The Maudsley Staging Method (MSM) assesses patients as having at least moderate refractory levels (MSM score ≥ 7);
* (6) Before randomization, the current antidepressant treatment regimen should be stable for at least 4 weeks, and the dosage used should not be lower than the prescribed range of drug use;
* (7) Having received education for 5 years or more;
* (8) Understand the experiment and sign an informed consent form.

Exclusion Criteria:

* (1) Meets the DSM-5 diagnostic criteria for other mental disorders, including schizophrenia spectrum disorders, bipolar and related disorders, neurodevelopmental disorders, neurocognitive disorders, or depression caused by substances and/or drugs, or depression caused by other medical issues;
* (2) Individuals with pacemakers, cochlear implants, or other metal foreign objects, as well as any electronic devices implanted in the body, contraindications for magnetic resonance imaging scans such as claustrophobia, and contraindications for rTMS treatment;
* (3) Concomitant history of epilepsy (with at least 2 non induced seizures with an interval of more than 24 hours, diagnosed with epilepsy syndrome, or having seizures within the past 12 months);
* (4) Individuals who have received modified electroconvulsive mECT, rTMS, or light therapy within 3 months;
* (5) Concomitant organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumors, etc.) and a history of severe brain injury;
* (6) Complicated with serious heart, liver, kidney diseases, diabetes and other serious physical diseases;
* (7) Women of childbearing age who are currently pregnant, breastfeeding, or planning or may become pregnant during the trial period;
* (8) Have a history of drug and alcohol abuse within the past year;
* (9) First degree relatives suffer from bipolar disorder;
* (10) There is a significant risk of suicide (the 10th item of the MADRS scale is ≥ 5 points);
* (11) Difficulty in verbal communication to the point of being unable to communicate normally, understand or follow instructions, and unable to cooperate with treatment and evaluation;
* (12) Currently participating in clinical trials of other drugs or physical therapies (such as deep brain stimulation (DBS), electroconvulsive therapy (ECT), rTMS);
* (13) The researchers believe it is not suitable to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from baseline to Immediate Post-treatment | Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from baseline to Immediate Post-treatment
  The Montgomery-Asberg Depression Rating Scale (MADRS) is a validated instrument stratifying the severity of depressive episodes in adults. The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression).

SECONDARY OUTCOMES:
Remission and response rates were estimated using Montgomery-Asberg Depression Rating Scale(MADRS) | Baseline, Day 21 (Immediate Post-treatment)
  The response is defined as a symptom improvement of ≥50% and remission is defined as a score ≤10 on MADRS
Remission and response rates were estimated using Hamilton Depression Rating Scale (HAMD-17) | Baseline, Day 21 (Immediate Post-treatment)
  The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The HAMD-17 version consists of 17 items，and has an overall score ranging from 0 (no depression) to 52 (worst depression). Higher scores represent higher depression severity. The response is defined as a symptom improvement of ≥50% and remission is defined as a score ≤7 on HAMD-17
Changes in the MADRS from baseline to each visit | Baseline, Day 21 (Immediate Post-treatment), 3-week Post-treatment, 9-week, and 6-month Post-treatment
  The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression). Higher scores represent higher depression severity.
Changes in the HAMD-17 from baseline to each visit | Baseline, Day 21 (Immediate Post-treatment), 3-week Post-treatment, 9-week Post-treatment
  The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The HAMD-17 version consists of 17 items，and has an overall score ranging from 0 (no depression) to 52 (worst depression). Higher scores represent higher depression severity.
cognitive change in Digit Symbol Substitution Test (DSST) | Baseline, Day 21 (Immediate Post-treatment)
  Cognitive scores are measured using Chinese brief cognitive test (C-BCT), the DSST equires a subject to match symbols to numbers according to a key located on the top of the page
cognitive change in continuous performance test (CPT) | Baseline, Day 21 (Immediate Post-treatment)
  CPT from the C-BCT measures a person's sustained and selective attention
cognitive change in Trail-Making Test (TMT) | Baseline, Day 21 (Immediate Post-treatment)
  The TMT test from the C-BCT can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning
cognitive change in Digit Span Test (DST) | Baseline, Day 21 (Immediate Post-treatment)
  DST from the C-BCT is a measure of verbal short term and working memory that can be used in two formats, Forward Digit Span and Reverse Digit Span

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (5):
- China (5):
  - Hebei Mental Health Center, Hebei, Baoding
  - West China Hospital, Sichuan University, Chengdu
  - Inner Mongolia Mental Health Center, Hohhot
  - Shandong Daizhuang Hospital, Jining
  - The Second Affiliated Hospital of Xinxiang Medical University, Xinxiang